CLINICAL TRIAL: NCT02133300
Title: Neuromuscular Electrical Stimulation in Critically Ill Patients
Brief Title: NMES in Critically Ill Patients
Acronym: NESCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Johan Segers, M.Sc., KU Leuven
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: u0064027
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Critically Ill Patients With a Predicted Prolonged ICU Stay
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- electrical stimulation (Experimental): Compex 3 professional NMES for 60' per day
  Interventions: Other: electrical stimulation
- control (No Intervention)

INTERVENTIONS:
Other: electrical stimulation
  Arms: electrical stimulation

SUMMARY:
Critically ill patients with a predicted prolonged ICU stay will receive neuromuscular electrical stimulation (NMES) of one quadriceps muscle. Whether the dominant or non-dominant side will be stimulated is chosen randomly by using opaque sealed envelopes. The patients will receive electrical stimulation for 1h for 7 consecutive days. The stimulated and non-stimulated side will be compared for it's thickness (by using ultrasound imaging), muscle strength if the patients are awake and cooperative (using the medical research council scale and handheld dynamometry) and a muscle biopsy will be taken. As a primary outcome the investigators hypothesize that electrical stimulation will preserve muscle mass with respect to the non-stimulated quadriceps. As secondary outcomes the investigators hypothesize that electrical stimulation can reduce muscle strength loss and leads to a better protein balance and thicker muscle fibers in the stimulated quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* All adult ICU patients with a predicted prolonged ICU stay

Exclusion Criteria:

* Preexisting neuromuscular disease, polyneuropathy or myopathy (e.g. Guillain-Barré, myasthenia gravis, Amyotrophic Lateral Sclerosis, paraplegia, multiple sclerosis, …)
* Receiving neuromuscular blocking agents
* Musculoskeletal conditions of the pelvis and/or lower limb (e.g. fractures, skin disease )
* Focal neurological conditions of the pelvis and/or lower limb
* Skin disease (e.g. burns)
* Presence of a pace-maker or defibrillator
* Hemodynamic or Respiratory Instability, active cardiac ischemia
* High fever (>39°)
* Pregnancy
* Brain death
* Intracranial pressure >20 mmHg
* An anticipated fatal outcome
* Psychiatric disorders or severe agitation
* Re-admission to the ICU

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | pre-intervention period
  Ultrasound measure in cm
Muscle thickness | post intervention period
  Ultrasound measure in cm

SECONDARY OUTCOMES:
Muscle strength (MRC & HHD) | pre intervention period
  MRC: scale HHD: MicroFet, in kg Force
Muscle fiber thickness | post intervention period
  biopsy using Bergström-Stille 5mm needles
Muscle strength (MRC & HHD) | post intervention period
  MRC: scale HHD: MicroFET, in kg Force
Protein balance | post intervention
  biopsy using Bergström-Stille 5mm needles

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Segers J, Vanhorebeek I, Langer D, Charususin N, Wei W, Frickx B, Demeyere I, Clerckx B, Casaer M, Derese I, Derde S, Pauwels L, Van den Berghe G, Hermans G, Gosselink R. Early neuromuscular electrical stimulation reduces the loss of muscle mass in critically ill patients - A within subject randomized controlled trial. J Crit Care. 2021 Apr;62:65-71. doi: 10.1016/j.jcrc.2020.11.018. Epub 2020 Nov 28. PMID 33285371